CLINICAL TRIAL: NCT00587210
Title: Evaluation of a New Oral Contrast Agent for MR Enterography in the Assessment of Crohn Disease in the Small Bowel
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeff Fidler, Professor of Radiology College of Medicine, Mayo Clinic
Other Study IDs: 381-04
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected or known Crohn Disease: Suspected or known Crohn Disease

SUMMARY:
The purpose of this study is to assess the exam quality and accuracy of MR using a new oral contrast agent for the evaluation of Crohn Disease in the small bowel.

DETAILED DESCRIPTION:
Crohn Disease is an inflammatory condition that involves the small bowel. Patients usually undergo multiple imaging exams in the diagnosis and surveillance of the disease. CT has been shown to have excellent results for detecting active inflammation. In the United States MR has lagged behind CT in utilization for imaging the small bowel. An advantage of MR over CT is the lack of radiation exposure to the patient. A new oral contrast agent is available that provides good distension of the small bowel and allows improved identification of active inflammation. The purpose of this study is to compare the accuracy of MR to CT using this new oral contrast agent and to assess exam quality.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected Crohn Disease
* Undergoing colonoscopy and CT enterography

Exclusion Criteria:

* Contraindication to MR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastroenteroloy Clinic; Inflammatory Bowel Disease Clinic
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2004-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
exam quality | one time point

CONTACTS AND LOCATIONS:
Overall Officials: Jeff L Fidler, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No